CLINICAL TRIAL: NCT01231100
Title: Effects of Hand-carried Ultrasound Echocardiography by Hospitalists Among Inpatients Referred for Standard Echocardiography: a Randomized Trial
Brief Title: Hand-carried Ultrasound Echocardiography in the Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook County Health (Other Government)
Responsible Party: Principal Investigator, Pamela Gonzalez Sr Director Clinical Research Office, Dir Clinical Research, Cook County Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCUE2
Record Dates: First submitted 2010-10-27; First posted 2010-11-01 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Adult Inpatients Referred for Standard Echocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HCUE-guided care (Experimental): Hand-carried ultrasound echocardiography
  Interventions: Other: HCUE-guided care
- Standard care (No Intervention)

INTERVENTIONS:
Other: HCUE-guided care — Care directed by hand-carried ultrasound echocardiography
  Arms: HCUE-guided care

SUMMARY:
The purpose of this study is to investigate whether or not care guided by hospitalists equipped with hand-carried ultrasound echocardiography reduces the length of stay of general medicine inpatients who were referred for standard echocardiography.

DETAILED DESCRIPTION:
This was an unblinded, parallel-group, superiority trial that randomized participants in a balanced (1:1) allocation ratio. We made no changes to our protocol after we began enrollment. Nor did we conduct any interim analyses. Each morning of the study period, including weekends and holidays, investigators listed all consecutive patients who were newly referred for SE by participating hospitalists. After hospitalists completed their initial evaluation of each patient, which included a history, physical exam, and review of medical records, investigators asked them to choose their indications for SE from a closed list. Given these indications, investigators then asked if HCUE could help them to assess their patients; if not, investigators excluded such patients. Finally, hospitalists were asked for their current management plans, which included medication regimens, diagnostic tests, specialty consultations, and timing of hospital discharge. If hospitalists remained masked to any preliminary SE results, investigators assigned participants who gave written informed consent to an intervention group. We used a computer-generated list of random numbers for the allocation sequence, and we concealed the sequence in an on-site computer system that only released allocations to investigators after they entered participant identifiers.

Hospitalists either awaited SE results for participants randomized to usual care or they performed HCUE for participants randomized to HCUE-guided care. Hospitalists performed HCUE with a MicroMaxx 3.4 hand-carried ultrasound machine equipped with a cardiology software package and a 1 to 5 MHz P17 cardiac transducer (Sonosite, Inc., Bothell, WA). The details of the HCUE protocol are described elsewhere. In brief, without assistance from nursing staff, hospitalists positioned participants on standard hospital beds and recorded 7 best-quality images up to 6 seconds in duration. Then hospitalists replayed the images for immediate interpretation. They made linear measurements with a caliper held directly to the ultrasound monitor and translated them into qualitative assessments based on simplified standard values.

The primary outcome was the length of stay on the short stay unit or general medicine ward service of the referring hospitalist. The duration began when the patient was admitted to the hospitalist service and ended when the patient was discharged home or transferred to a different service in the hospital. We chose this duration, rather than the length of stay of the entire hospitalization, because we wanted the primary outcome to reflect how HCUE affected hospitalists' management decisions in the hospital, including the transfer of participants to other services.

ELIGIBILITY:
Inclusion Criteria:

* general medicine inpatients 18 years or older who were referred for inpatient standard echocardiography by hospitalists trained in hand-carried ultrasound echocardiography

Exclusion Criteria:

* referring hospitalist not being masked to standard echocardiography results and determination by the referring hospitalist that hand-carried ultrasound echocardiography was unlikely to help given the indications for standard echocardiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 453 (Actual)
Dates: Start 2008-07; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Length of stay on referring hospitalist's service | From date of randomization until the date of tranfer off the referring hospitalist's service (including death from any cause), assessed up to 1 month after admission to the hospitalist's service.
  The length of stay begins when the patient arrives on the referring hospitalist's service and end when the patient leaves the referring hospitalist's service.

SECONDARY OUTCOMES:
Unplanned repeat visit to hospital or emergency department | 30 days after discharge from hospital
  From date of discharge from the hospital and from the referring hospitalist's service until an unplanned visit back to our hospital or emergency department, assessed up to 30 days after discharge.
Time to performance of standard echocardiography. | From time of admission until the time of performance of standard echocardiography, assessed up to 1 week after time of admission.

CONTACTS AND LOCATIONS:
Overall Officials: Brian P Lucas, MD MS FHM, Principal Investigator — Stroger Hospital of Cook County
Locations (1):
- Stroger Hospital of Cook County, Chicago, Illinois, United States